CLINICAL TRIAL: NCT04383067
Title: A Phase 2, Single-Center, Open Label Study of Autologous, Adoptive Cell Therapy Following a Reduced Intensity, Non-myeloablative, Lymphodepleting Induction Regimen in Metastatic Urothelial Carcinoma Patients
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Principal Investigator, Dr. Ronnie Shapira, Director , The Ella Lemelbaum Institute of Immuno-Oncology, Principal Investigator, Associate Professor of Immunology, Sheba Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHEBA-19-6407-RS-TIL TCC
Record Dates: First submitted 2020-05-03; First posted 2020-05-11 (Actual); Last update posted 2021-02-11 (Actual); Status verified 2020-05

CONDITIONS: Metastatic Urothelial Carcinoma
Keywords: Urothelial cancer; Tumor infiltrating lymphocytes; Cellular therapy
MeSH Terms: conditions — Carcinoma, Transitional Cell | interventions — aldesleukin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Tumor Infiltrating Lymphocytes (TIL) (Experimental)
  Interventions: Procedure: Tumor Infiltrating Lymphocytes (TIL); Drug: Proleukin

INTERVENTIONS:
Procedure: Tumor Infiltrating Lymphocytes (TIL) — Patient with metastatic urothelial carcinoma will undergo a autologous lymphocyte transplantation. Patient will undergo surgery to remove either the primary tumor or a tumor metastasis. The cells collected in this surgey will be cultured and reintroduced to the patient. Following the cell infusion, patient will receive a high-dose bolus of IL-2.
Drug: Proleukin — high-dose (720,000 IU/kg) IL-2 will be administered every 8 hours, to tolerance. A maximum of 10 doses will be administered

SUMMARY:
An autologous, Adoptive Cell Therapy Following a Reduced Intensity, Non-myeloablative, Lymphodepleting Induction Regimen in Metastatic Urothelial Carcinoma Patients.

DETAILED DESCRIPTION:
This is a phase II single-center study of Tumor Infiltrating Lymphocytes (TIL) in urothelial carcinoma patients who failed at least one line of platinum based chemotherapy and one line of immunotherapy of targeted therapy.

Patients will undergo a baseline evaluation including imaging, blood and urine samples, EVG and physical examination to confirm suitability for the study.

Eligible patients will undergo surgery to collect a tumor sample for TIL culturing.

Patients will receive an autologus TIL infusion once the cells have been properly cultured.

Following the infusion, patients will receive a high dose of IL-2.

Following the intervention, patients will be monitored to evaluate study endpoints.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed Urothelial Carcinoma
2. Progressed on first line platinum-based chemotherapy and on second line immunotherapy or targeted therapy (FGFR inhibitor)
3. Measurable metastatic Urothelial Carcinoma with at least one lesion that is resectable for TIL generation.
4. Patients with one or more brain metastases less than 1 cm each, and any patients with 1 or 2 brain metastases greater than 1 cm must have been treated and stable for 4 weeks.
5. Greater than or equal to 18 years of age.
6. Willing to practice birth control from the start of chemotherapy until 120 days after release from the hospital.
7. Life expectancy of greater than three months
8. Willing to sign a durable power of attorney
9. Able to understand and sign the Informed Consent Document
10. Clinical performance status of ECOG 0 or 1
11. Hematology:

    * Absolute neutrophil count greater than 1000/mm3 without support of filgrastim
    * Normal WBC ( > 3000/mm3).
    * Hemoglobin greater than 8.0 g/dL
    * Platelet count greater than 100,000/mm3
12. Serology:

    * Seronegative for HIV antibody. (The experimental treatment being evaluated in this protocol depends on an intact immune system. Patients who are HIV seropositive can have decreased immune competence and thus can be less responsive to the experimental treatment and more susceptible to its toxicities.)
    * Seronegative for Hepatitis B or Hepatitis C. (patients who recovered from previous infection and have no detected HBSAg or HCV RNA are allowed).
13. Chemistry:

    * Serum ALT/AST less than three times the upper limit of normal (ULN).
    * Serum creatinine less than or equal to 1.6 mg/dL
    * Total bilirubin no more than x1.5 times the ULN, except in patients with Gilbert's Syndrome who must have a total bilirubin less than 3 mg/dL.
14. Negative pregnancy test in women of child bearing potential because of the potentially dangerous effects of the preparative chemotherapy on the fetus.
15. More than four weeks must have elapsed since any prior systemic therapy at the time the patient receives the preparative regimen, and patients' toxicities must have recovered to a grade 1 or less (except for toxicities such as alopecia or vitiligo). Patients may have undergone minor surgical procedures with the past 3 weeks, as long as all toxicities have recovered to grade 1 or less.

Exclusion Criteria:

1. Upper tract Urothelial Carcinoma
2. History of nephrectomy
3. Women of child-bearing potential who are pregnant or breastfeeding because of the potentially dangerous effects of the non-myeloablative, lymphodepleting induction regimen on the fetus or infant.
4. Systemic steroid therapy required (patients that require replacement therapy for adrenal insufficiency may be enrolled if steroid treatment dose do not exceed 10 mg of prednisone or equivalent).
5. Active systemic infections, coagulation disorders or other active major medical illnesses of the cardiovascular, respiratory or immune system, as evidenced by a positive stress thallium or comparable test, myocardial infarction, cardiac arrhythmias, obstructive or restrictive pulmonary disease.
6. Any form of primary immunodeficiency (such as Severe Combined Immunodeficiency Disease and AIDS).
7. Opportunistic infections (the experimental treatment being evaluated in this protocol depends on an intact immune system. Patients who have decreased immune competence may be less responsive to the experimental treatment and more susceptible to its toxicities.)
8. History of severe immediate hypersensitivity reaction to any of the agents used in this study, including history of an anaphylactic reaction to penicillin or gentamicin
9. History of coronary revascularization or ischemic heart disease.
10. Any patient known to have an LVEF less than or equal to 50%.
11. Documented LVEF of less than or equal to 50% tested in patients with clinically significant atrial and/or ventricular arrhythmias including but not limited to: atrial fibrillation, ventricular tachycardia, second- or third-degree heart block
12. Documented FEV1 and DLCO (relative to predicted) less than or equal to 60%

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2020-05-12 (Actual); Primary Completion 2022-06-01 (Estimated); Study Completion 2023-06-01 (Estimated)

PRIMARY OUTCOMES:
Efficacy endpoint Objective Tumor response according to RECICT 1.1 | 3 Years
  The primary efficacy endpoint is defined as at least a 20% clinical benefit expressed as the sum of CR+PR+SD (each of these parameters defined as persisting for at least for 12 weeks).
Safety endpoint Assess Adverse Events using CTCAE V4.03 during treatment and FU | 3 Years
  The primary safety endpoint of the study is to evaluate the overall toxicity profile of the ACT procedure, with an emphasis on the side effects of the reduced intensity, non-myeloablative, lymphodepleting induction regimen.

SECONDARY OUTCOMES:
Overall Survival | 3 Years
  Overall Survival (OS) according to RECICT 1.1
Progression-Free Survival | 3 Years
  Progression-Free Survival (PFS) according to RECICT 1.1
Quality of Life (QoL) Assessment | 3 Years
  Assessment of QoL using disease specific modules of the EORTC QLQ-C30 (version 3.0)

OTHER OUTCOMES:
Tissue markers assessment | 3 Years
  Tissue markers such as protein expression
Blood Bio-markers assessment | 3 Years
  Blood Bio-markers, including Circulating factors and peripheral blood mononuclear cell phenotype and function

CONTACTS AND LOCATIONS:
Locations (1):
- Sheba Medical Center, Ramat Gan, Israel